CLINICAL TRIAL: NCT03836911
Title: Effects of a Serious Game Based Exercise Program on the Functional Autonomy in Older Adults Living in Nursing Homes : SERIOUS AUTONOMY
Brief Title: Effects of a Serious Game With Elderly People
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Sanitary context (COVID19)
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: RECHMPL18_0006; NCT03694795 (obsolete NCT alias)
Record Dates: First submitted 2018-09-17; First posted 2019-02-11 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2025-01

CONDITIONS: Functional Autonomy
Keywords: Institutionalized olders adults; SERIOUS GAME

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- serious game (Active Comparator): the effect on physical performance of a personalized, 12-weeks rehabilitation program using a serious game
  Interventions: Other: serious game
- Classic program (Other): the effect on physical performance of a personalized, 12-weeks rehabilitation program using a classical exercise program in older subjects living in a nursing home
  Interventions: Other: classic program

INTERVENTIONS:
Other: serious game — Effect of serious game on elderly in comparison of the physical activity adapted meeting
  Arms: serious game
Other: classic program — Effect of serious game on elderly in comparison of the physical activity adapted meeting
  Arms: Classic program

SUMMARY:
Assessment of the effect of a 12 weeks serious game based exercises program on physical performance in older adults living in nursing homes, in comparison with a control group that benefits from a classical exercise training program including balance, muscle strengthening and walking exercises with the same duration.

DETAILED DESCRIPTION:
Recent reviews of the literature have shown that exergames may have interest in balance rehabilitation, physical performance maintenance, and fall prevention in community dwelling older adults with neurodegenerative disease or at risk of fall. These reviews also show however that classical exergames are not adapted for rehabilitation of patients with functional limitations, which could explain their relatively moderate benefits in those patients.

To overcome this lack, a serious game has been co-developed with medical to be adapted to the specific needs and characteristics of nursing home residents In this study , the investigators propose to compare the effects on physical performance, falls incidence, and quality of life of a 12-weeks serious game based exercise program and a classical exercises program

ELIGIBILITY:
Inclusion Criteria:

* older adults aged 65 and over, living in nursing homes and able to walk without technical assistance and sign an informed consent.

Exclusion Criteria:

* subjects with cognitive impairments (MMSE < 14) or with conditions that contra-indicate the involvement in a rehabilitation program for medical or ethics reasons; subjects with a history of seizure.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 136 (Actual)
Dates: Start 2019-02-28 (Actual); Primary Completion 2022-10-28 (Actual); Study Completion 2022-10-28 (Actual)

PRIMARY OUTCOMES:
Short Physical Performance Baterry (SPPB) | 3 months
  Short Physical Performance Baterry (SPPB) at baseline (T0) and at 3 months.The Short Physical Performance Battery (SPPB) is the sum of the scores on three criteria: the balance test, the walking speed test and the chair lift test. This test makes it possible to evaluate the physical performance of an individual.

SECONDARY OUTCOMES:
Short Physical Performance Baterry (SPPB) | 6 months
  SPPB score at 6 months.The Short Physical Performance Battery (SPPB) is the sum of the scores on three criteria: the balance test, the walking speed test and the chair lift test. This test makes it possible to evaluate the physical performance of an individual.
incidence of fall | 3 months
  incidence of fall
incidence of fall | 6 months
  incidence of fall
Balance | at baseline (T0)
  Timed Up and Go Test, Tinetti Test and unipodal standing in simple and dual-task
Balance | 3 months
  Timed Up and Go Test, Tinetti Test and unipodal standing in simple and dual-task
Cognition | At inclusion
  Mini Mental State Examination
Cognition | 3 months
  Mini Mental State Examination
Satisfaction evaluation | At inclusion
  Lickert Scale at inclusion.A Likert scale is a psychometric tool to measure an attitude in individuals.The scale contains for each item a graduation generally comprising five or seven answer choices that qualify the degree of agreement
Satisfaction evaluation | 3 months
  Lickert Scale at inclusion.A Likert scale is a psychometric tool to measure an attitude in individuals.The scale contains for each item a graduation generally comprising five or seven answer choices that qualify the degree of agreement
Evaluation of the quality of life | At inclusion
  SF12 questionnaire
Evaluation of the quality of life | 3 months
  SF12 questionnaire

CONTACTS AND LOCATIONS:
Locations (15):
- France (15):
  - EHPAD Les Aigueillières, Montferrier-sur-Lez
  - EHPAD Françoise Gauffier CCAS de Montpellier, Montpellier
  - Ehpad Maison de Famille, Montpellier
  - EHPAD Pierre Laroque CCAS de Montpellier, Montpellier
  - EHPAD Le Barry, Muret
  - EHPAD Marie-Antoinette, Muret
  - EHPAD Résidence La Camargue, Nimes (Groue Orpéa), Nîmes
  - EHPAD Résidence Château Notre Dame (Groupe Orpéa), Parignargues
  - EHPAD Belleviste, Saint-Gély-du-Fesc
  - EHPAD Caroline Baron, Toulouse
  - Ehpad La Cotonniere, Toulouse
  - EHPAD LA houlette, Toulouse
  - Ehpad Le Bois Vert, Toulouse
  - Ehpad Pastelliere, Toulouse
  - EHPAD Le Grand Marquisat, Tournefeuille

IPD SHARING:
Plan to Share IPD: No